CLINICAL TRIAL: NCT03889197
Title: Physiologic Approach to Sodium Supplementation in Premature Infants
Acronym: Salt to Grow
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Gregory M Sokol, Professor of Clinical Pediatrics, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1902815407
Record Dates: First submitted 2019-03-18; First posted 2019-03-26 (Actual); Results first posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-08

CONDITIONS: Postnatal Growth Disorder
Keywords: Postnatal Growth Disorder; Growth and development

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data entered as group A and B.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Standard of care sodium supplementation as directed by the medical care team
- Sodium supplementation algorithm (Active Comparator): Beginning on the 14th -16th postnatal day and continuing until 36 weeks postmenstrual age, infants randomized to the algorithm will have a spot urine sodium concentration determined every two weeks and sodium supplementation provided according to the algorithm.
  Interventions: Drug: Sodium supplementation guided by urine sodium concentration algorithm

INTERVENTIONS:
Drug: Sodium supplementation guided by urine sodium concentration algorithm — 4 mEq/kg/d sodium added the first time urine [Na] below threshold; for each subsequent time urine [Na] below threshold, add additional 2 mEq/kg/d.
  Arms: Sodium supplementation algorithm

SUMMARY:
Postnatal growth failure occurs in up to 50% of very low birth weight (VLBW, <1500 grams at birth) infants as assessed by discharge weight. This study will evaluate if a sodium supplementation algorithm guided by spot urine sodium measurements can improve postnatal growth.

DETAILED DESCRIPTION:
Postnatal growth failure is a significant morbidity in very low birth weight (VLBW, <1500 grams at birth) infants. Efforts to promote growth and optimize nutritional support have included earlier initiation of parenteral nutrition and increased caloric and protein administration. While these advances in nutritional practices have resulted in improved growth, up to 50% of VLBW infants continue to experience postnatal growth failure (defined as discharge weight <10th percentile by Fenton growth charts) and over 25% experience severe postnatal growth failure (<3rd percentile). Current nutritional recommendations for sodium provision to preterm infants is 3-5 mEq/kg/d and fails to take into account the degree of renal immaturity present in extremely preterm infants. The investigators hypothesize that the sodium supplementation algorithm will improve in-hospital somatic growth (weight, length, and head circumference) between 2 weeks of postnatal age and 36 weeks postmenstrual age over current sodium replacement practices. The algorithm will be evaluated in a prospective, pragmatic, randomized trial. Infants in the sodium supplementation algorithm group will have a spot urine sodium concentration determined every two weeks beginning on the 14th postnatal day and continuing until 36 weeks postmenstrual age with sodium supplementation provided according to the algorithm.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with gestational age 25 0/7 - 29 6/7 at birth
2. Birth weight ≥ 500 grams
3. Admitted within the 1st week of life
4. < 17 days of age at time of enrollment

Exclusion Criteria:

1. Infants admitted after the 1st week of life
2. Major congenital anomalies
3. Structural genitourinary abnormality
4. Renal dysfunction (serum creatinine > 1.0 mg/dl or an increase of ≥ 0.3 mg/dl between the 2 most recent consecutive measurements) immediately prior to the initiation of study procedures.
5. Diuretic use less than 48 hours prior to initiation of study procedures
6. Infant with an ostomy (infants receiving an ostomy after study entry will be withdrawn)
7. Infant with a diagnosis or suspicion of diabetes insipidus

Ages: 7 Days to 16 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Sokol, MD, Principal Investigator — Indiana University; Jeffrey L Segar, MD, Principal Investigator — Medical College Wisconsin
Locations (3):
- United States (3):
  - Indiana University Health North, Carmel, Indiana
  - Riley Hospital for Children at IU Health, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segar DE, Segar EK, Harshman LA, Dagle JM, Carlson SJ, Segar JL. Physiological Approach to Sodium Supplementation in Preterm Infants. Am J Perinatol. 2018 Aug;35(10):994-1000. doi: 10.1055/s-0038-1632366. Epub 2018 Feb 27. PMID 29486497

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 3 level III NICUs and 1 level IV NICU within an academic health care system between July 2019 and August 2023.
Pre-assignment Details: Of the 385 infants screened for eligibility, 260 met inclusion/exclusion criteria, and 90 provided informed consent.
Period: Overall Study
Arm/Group | Control | Sodium Supplementation Algorithm
Started | 45 | 45
Completed | 43 | 43
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1
Not completed — met exclusion criteria | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Sodium Supplementation Algorithm | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 28.00 (1.44) | 27.87 (1.36) | 27.93 (1.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 24 | 48
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 34 | 38 | 72
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 26 | 30 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43 | 43 | 86
Singleton [Count of Participants; unit: Participants] — A pregnancy with one baby or fetus.
  Participants | 30 | 38 | 68
Inborn [Count of Participants; unit: Participants] — Infant born at the study center.
  Participants | 40 | 41 | 81
Birth Weight [Mean (Standard Deviation); unit: kilograms] | 1.14 (0.24) | 1.13 (0.28) | 1.13 (0.26)
Birth Weight z-score [Mean (Standard Deviation); unit: Z-score] — The Z-score (standard score) provides a measure of how many standard deviations above or below the population mean the infant birth weight is. A Z-score of 0 represents the population mean. A positive z-score would indicate better growth.
  Z-score | 0.45 (0.93) | 0.24 (0.96) | 0.35 (0.94)
Birth Length [Mean (Standard Deviation); unit: cm] — Population: Data was missing for 1 participant in the control arm because it was not collected.
  cm
    number analyzed (Participants) | 42 | 43 | 85
    (all) | 36.05 (3.04) | 36.29 (3.03) | 36.17 (3.02)
Birth Length z-score [Mean (Standard Deviation); unit: Z-score] — The Z-score (standard score) provides a measure of how many standard deviations above or below the population mean the infant birth length is. A Z-score of 0 represents the population mean. A positive z-score would indicate better growth. Population: Data was missing for 1 participant in the control arm because it was not collected.
  Z-score
    number analyzed (Participants) | 42 | 43 | 85
    (all) | 0.04 (1.10) | -0.11 (1.63) | -0.03 (1.39)
Birth Head Circumference [Mean (Standard Deviation); unit: cm] | 25.70 (1.82) | 25.16 (2.12) | 25.43 (1.98)
Birth Head Circumference z-score [Mean (Standard Deviation); unit: Z-score] — The Z-score (standard score) provides a measure of how many standard deviations above or below the population mean the infant birth head circumference is. A Z-score of 0 represents the population mean. A positive z-score would indicate better growth.
  Z-score | 0.25 (0.99) | -0.16 (1.18) | 0.05 (1.10)
Small for Gestational Age (< 3rd percentile) [Number; unit: participants] — The Fenton growth chart is a reference chart based on size at birth by gestational age. The 50th percentile would be the mean weight for gestational age. An infant < 3rd percentile would be a severely growth restricted infant.
  participants | 2 | 2 | 4
Received Antenatal glucocorticoids [Count of Participants; unit: Participants] | 34 | 40 | 74
Cesarian Delivery [Count of Participants; unit: Participants] | 34 | 31 | 65
Apgar Score at 1 minute [Mean (Standard Deviation); unit: scores on a scale] — APGAR score = Appearance, Pulse, Grimace, Activity, Respiration. A value of 0-2 is assigned for each component; providing a range of scores from 0-10. The 1-minute score describes how the infant tolerated the birthing process. Higher scores are better.
  scores on a scale | 4.51 (2.29) | 4.77 (2.11) | 4.64 (2.20)
Apgar Score at 5 minutes [Mean (Standard Deviation); unit: scores on a scale] — APGAR score = Appearance, Pulse, Grimace, Activity, Respiration. A value of 0-2 is assigned for each component; providing a range of scores from 0-10. The 5-minute score describes how the infant is tolerating being outside of the mothers womb. Higher scores are better.
  scores on a scale | 6.53 (2.11) | 6.56 (1.59) | 6.55 (1.86)
Age at Randomization [Mean (Standard Deviation); unit: Days] — The "Age at Randomization" is the day of age each participant began study participation (intervention if so randomized) and is the starting point for growth assessment outcomes. Other characteristics at birth were included as baseline measures to provide general descriptors of newborn infants.
  Days | 14.35 (1.23) | 14.33 (1.23) | 14.34 (1.22)

OUTCOME MEASURES:

1. Primary Outcome: Change in Somatic Growth (Weight)
Description: Evaluated by the change in Z-score (standard score) provides a measure of how many standard deviations above or below the population mean the infant weight is. A Z-score of 0 represents the population mean. A positive z-score would indicate better growth.
Time Frame: between 2 weeks of age and 36 weeks post-menstrual age or transfer from the NICU (whichever occurs first).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
score on a scale | 0.04 (0.63) | 0.16 (0.41)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.162, Kruskal-Wallis

2. Primary Outcome: Change in Somatic Growth (Length)
Description: Evaluated by the change in Z-score (standard score) provides a measure of how many standard deviations above or below the population mean the infant length is. A Z-score of 0 represents the population mean. A positive z-score would indicate better growth.
Time Frame: between 2 weeks of age and 36 weeks post-menstrual age or transfer from the NICU (whichever occurs first).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
score on a scale | -0.34 (0.66) | -0.48 (0.48)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.242, Kruskal-Wallis

3. Primary Outcome: Change in Somatic Growth (Head Circumference)
Description: Evaluated by the change in Z-score (standard score) provides a measure of how many standard deviations above or below the population mean the infant head circumference is. A Z-score of 0 represents the population mean. A positive z-score would indicate better growth.
Time Frame: between 2 weeks of age and 36 weeks post-menstrual age or transfer from the NICU (whichever occurs first).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
score on a scale | 0.60 (0.88) | 0.54 (0.57)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.956, Kruskal-Wallis

4. Secondary Outcome: Change in Somatic Growth (Weight) at Discharge/Transfer
Description: as for outcome 1
Time Frame: between 2 weeks of age and discharge/transfer from hospital, up to 44 weeks post-menstrual age (whichever occurs first).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
score on a scale | 0.04 (0.80) | 0.24 (0.76)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.132, Kruskal-Wallis

5. Secondary Outcome: Change in Somatic Growth (Weight) at Discharge/Transfer
Description: evaluated by the change in kilograms
Time Frame: between 2 weeks of age and discharge/transfer from hospital, up to 44 weeks post-menstrual age (whichever occurs first).
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
kilograms | 2.00 (0.76) | 2.14 (0.82)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.445, Kruskal-Wallis

6. Secondary Outcome: Change in Somatic Growth (Length) at Discharge/Transfer
Description: as for outcome 2
Time Frame: between 2 weeks of age and discharge/transfer from the NICU or 44 weeks post-menstrual age (whichever occurs first)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
score on a scale | -0.39 (0.96) | 0.92 (8.56)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.746, Kruskal-Wallis

7. Secondary Outcome: Change in Somatic Growth (Head Circumference) at Discharge/Transfer
Description: as for outcome 3
Time Frame: between 2 weeks of age and discharge/transfer from the NICU or 44 weeks post-menstrual age (whichever occurs first)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
score on a scale | 1.03 (1.07) | 2.07 (7.39)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.979, Kruskal-Wallis

8. Secondary Outcome: Received Diuretic Therapy
Description: number of participants who received diuretic therapy
Time Frame: between 2 weeks of age and discharge/transfer from the NICU or 44 weeks post-menstrual age (whichever occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
Participants | 7 | 11
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.289, Chi-squared

9. Secondary Outcome: Duration of Mechanical Ventilation
Description: days on assisted ventilation
Time Frame: from birth to discharge/transfer from the NICU or 44 weeks post-menstrual age (whichever occurs first)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
Days | 12.60 (44.38) | 8.74 (16.08)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.940, Kruskal-Wallis

10. Secondary Outcome: Need for Supplemental Oxygen at Discharge
Description: supplemental oxygen requirement
Time Frame: assessed at discharge/transfer from the NICU or 44 weeks post-menstrual age (whichever occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
Participants | 7 | 13
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.126, Chi-squared

11. Secondary Outcome: Incidence and Severity of Bronchopulmonary Dysplasia (BPD)
Description: Jenson definition of bronchopulmonary dysplasia (BPD), rated 0 - 3; with 0 being no BPD and higher numbers being more severe disease
Time Frame: determined at 36 weeks post-menstrual age
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
Participants
  Grade 0 | 16 | 15
  Grade 1 | 11 | 10
  Grade 2 | 12 | 16
  Grade 3 | 4 | 2
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.738, Fisher Exact

12. Secondary Outcome: Retinopathy of Prematurity ≥ Stage 3
Description: Number of participants with Retinopathy of prematurity ≥ Stage 3 as diagnosed by examination of an Ophthalmologist finding abnormal retinal blood vessel growth with ridge formation or retinal detachment.
Time Frame: assessed at discharge/transfer from the NICU or 44 weeks post-menstrual age (whichever occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 43 | 43
Participants | 4 | 2
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.676, Fisher Exact

13. Secondary Outcome: Total Body Water
Description: Calculated by the doubly labeled water method in ml/kg
Time Frame: determined during participants 32nd post-menstrual week of life
Population: Samples not collected for 6 Control participants and 4 Sodium supplementation algorithm participants.
Measure: Mean (Standard Deviation); unit: ml/kg of water
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 37 | 39
ml/kg of water | 755.5 (41.4) | 756.2 (41.6)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.996, Kruskal-Wallis

14. Secondary Outcome: Energy Expenditure
Description: Calculated using the doubly labeled water method
Time Frame: determined during the participants 32nd post-menstrual week of life
Population: Samples were not collected for 2 Control participants and 1 Sodium supplementation algorithm participant.
Measure: Mean (Standard Deviation); unit: kcal/kg/d
Arm/Group | Control | Sodium Supplementation Algorithm
Number analyzed (Participants) | 41 | 42
kcal/kg/d | 61.6 (9.6) | 65.4 (9.8)
Statistical Analysis 1: Comparison: Control vs Sodium Supplementation Algorithm; Test type: Superiority; p = 0.095, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: from study intervention (~ 2 weeks of age) until 36 weeks post-menstrual age or participant discharged or transferred to another hospital (whichever occurred first).
Description: Extremely preterm infants commonly have multiple clinical complications and laboratory abnormalities associated with prematurity. Special clinical outcomes of interest are listed in secondary outcomes.
Arm/Group | Control | Sodium Supplementation Algorithm
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 3/43 | 2/43
Other Adverse Events (participants affected / at risk) | 5/43 | 9/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=43) | Sodium Supplementation Algorithm (N=43)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — serum sodium < 130
Edema/Anasarca (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — As per identified by care giver physical exam.
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) — As identified by clinician.
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (3) | 0 (0) — As identified by clinician.
post-NEC adhesions (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=43) | Sodium Supplementation Algorithm (N=43)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2) | 4 (4) — participants with 2 consecutive serum sodium levels greater than 145
Hyponatremia (Metabolism and nutrition disorders) | 5 (15) | 7 (14) — participants with 2 consecutive serum sodium measurements less than 135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-10-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT03889197/Prot_SAP_ICF_000.pdf